CLINICAL TRIAL: NCT04423120
Title: A Single Arm, Multicenter, Prospective, Clinical Study on a Novel Minimally Invasive Posterior Sacroiliac Fusion Device
Brief Title: Clinical Study on a Novel Minimally Invasive Posterior Sacroiliac Fusion Device
Status: Completed | Type: Observational
Sponsor: PainTEQ, LLC (Industry)
Collaborators: Pacific Research Institute (Network)
Responsible Party: Sponsor
Other Study IDs: SECURE
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PainTEQ study is a prospective, multi-site, prospective, single arm study intended to collect clinical data outcomes data associated with the treatment of sacroiliac disease with the LinQ fusion procedure. Data will be collected using self-report measures including the visual analog scale (VAS) for pain assessment where the participant is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. Other self-report questionnaires will be administered including the Oswestry Disablity Index (ODI) to measure low-back pain and disability, and the Patient-Reported Outcomes Measurement Information System 29 (PROMIS 29) to measure physical, mental, and social health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70
* Patient has lower back pain for >6 months inadequately responsive to conservative care
* Patient has at least 3 of 4 physical examination maneuvers specific for the SI joint (FABER, Gaenslen test, Stork/Gillete, and Yoman)
* Patient has improvement in lower back pain numeric rating scale (NRS) of at least 50% after injection of local anesthetic into affected SI joint(s) with confirmed arthrogram, within 30-60 min from injection
* Degenerative sacroiliitis as SIJ mediated in in the context of either radiographic evidence of SIJ degeneration, evident on computed tomography or Xrays or a history of prior lumbar fusion.
* SIJ disruption was defined in the study of as SIJ mediated pain in the context of asymmetric widening of SIJ on CT or Xrays or the presence of significant contrast leakage during diagnostic SIJ block
* Baseline Oswestry Disability Index (ODI) score of at least 30%
* Baseline Low back/buttock pain score of at least 50 on 0-100 mm visual analog scale
* Patient has signed study-specific informed consent form
* Patient has the necessary mental capacity to consent and participate and is physically able to comply with study protocol requirements
* Patient has medical insurance that covers this standard of care procedure and all other anticipated and unanticipated procedure related care.
* Patient's physician has decided that the best treatment for the patient's sacro-iliac disease is the LinQ system and the patient has agreed to the treatment.

Exclusion Criteria:

* Inability to confirm that the pain is arising from the sacroiliac joint
* Current severe back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, lumbar radicular pain, and lumbar vertebral body fracture
* SIJ pain secondary to inflammatory conditions, Other known sacroiliac pathology such as: Sacral dysplasia, Inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondylo-arthropathy), Tumor, Infection, Acute fracture, and Crystal arthropathy.
* Radicular pain extending beyond the buttock ≥ 30mm on VAS
* Has complete resolution of pain from the diagnostic SIJ injection lasting 30 days or more
* Has had an injection with corticosteroid into the index SIJ within the last 90 days
* Has had any neuraxial injection with corticosteroid within the last 90 days
* Has greater than 50% pain relief from diagnostic medial branch blocks at the L4/5 and/or L5/S1 levels
* Has had a sacral radiofrequency ablation within the last 6 months
* History of any hardware placement within the sacrum or sacroiliac joint
* History of coccydynia or coccygectomy
* Clinical diagnosis of discogenic pain at L4/5 and/or L5/S1
* History of endometriosis or pudendal neuralgia
* History of recent (<1 year) major trauma to pelvis
* Chronic rheumatologic condition (e.g., rheumatoid arthritis)
* Any condition or anatomy that makes treatment with the Linq Implant System infeasible
* Use of medications known to have detrimental effects on bone quality and soft-tissue healing (metabolic bone disease, induced or idiopathic)
* Prominent neurologic condition that would interfere with physical therapy
* Current local or systemic infection that raises the risk of surgery
* Patient currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation.
* Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation
* Patient with insurance coverage that does not cover the SI fusion*
* Implanted intrathecal pain pump

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will come from the existing patient population of the investigators in each individual practice.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline VAS Sacroiliac Joint (SIJ) pain by at least 20 millimeters | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  A subject was considered a success if all of the following criteria were met
  1. Change from baseline VAS SIJ pain by at least 20 mm (Binary success failure composite end point) VAS is a vertical scale, where a higher score depicts more pain (100 mm maximum) and a lower scale depicts less pain (0 mm minimum)
Absence of device related serious adverse events | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  A subject was considered a success if all of the following criteria were met
  2. Absence of device related serious adverse events, (Binary success failure composite end point)
Absence of neurological worsening related to the lumbosacral nerve roots | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  A subject was considered a success if all of the following criteria were met
  3. Absence of neurological worsening related to the lumbosacral nerve roots, (Binary success failure composite end point)
Absence of surgical reintervention (removal, revision reoperation or supplemental fixation) for SIJ pain | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  A subject was considered a success if all of the following criteria were met
  4. Absence of surgical reintervention (removal, revision reoperation or supplemental fixation) for SIJ pain (Binary success failure composite end point)

SECONDARY OUTCOMES:
Change in VAS | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  1. Change in baseline in VAS from baseline at 6 months
Change in ODI | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  2. Change in Oswestry Disability Index at 6 months follow up ODI assesses disability and has 10 sections, each with a point range from 0 (minimum) to 5 (maximum). A higher score translates to a higher percentage, meaning more disability (100% maximum). A lower score translates to a lower percentage, meaning less disability (0% minimum).
Change in PROMIS29 | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  3. Change in PROMIS-29 at 6 months follow up. PROMIS 29 assesses pain intensity using a 0-10 numeric rating scale (11 point scale), where a higher score equates to more pain. Other health domains are scored using a Likert scale, where higher scores represent more of the specific domain being measured.
Change in Patient Global Impression of Change (PGIC) | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  4. Change in Patient Satisfaction with PGIC PGIC is on a 7 point scale that depicts a patient's rating on their overall improvement. A lower score translates to a profound improvement and a higher score translates to a salvage improvement.
Change in Morphine milligram equivalent | Comparisons will be done prior to baseline visit and 7-14 days post surgery, 1 month, 3 month, 6 month, and 12 month visits.
  5. Change in MME usage at all time points

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Calodeny, MD, Principal Investigator — Precision Spine Care
Locations (1):
- Precision Spine Care, Tyler, Texas, United States

REFERENCES:
- [Result] Calodney A, Azeem N, Buchanan P, Skaribas I, Antony A, Kim C, Girardi G, Vu C, Bovinet C, Vogel R, Li S, Jassal N, Josephson Y, Lubenow T, Lam CM, Deer TR. Safety, Efficacy, and Durability of Outcomes: Results from SECURE: A Single Arm, Multicenter, Prospective, Clinical Study on a Minimally Invasive Posterior Sacroiliac Fusion Allograft Implant. J Pain Res. 2024 Mar 20;17:1209-1222. doi: 10.2147/JPR.S458334. eCollection 2024. PMID 38524688

DOCUMENTS (1):
  • Study Protocol (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT04423120/Prot_000.pdf